CLINICAL TRIAL: NCT05674448
Title: An Open-label Phase IIa Study to Evaluate the Antiviral Effect and Safety of HH-003 Injection in Subjects With Chronic Hepatitis B and D Co-infection
Brief Title: A Study to Evaluate the Antiviral Activity and Safety of HH-003 Injection in Subjects With Chronic Hepatitis B and Hepatitis D Co-infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: During the study, the sponsor adjusted the overall clinical development strategy, decided to terminate the enrollment in advance after discussion with the lead investigator.
Sponsor: Huahui Health (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HH003-201
Record Dates: First submitted 2022-12-30; First posted 2023-01-06 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2022-12

CONDITIONS: Chronic Hepatitis B and Hepatitis D Co-infection
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HH-003 20mg/kg (Experimental): HH-003 20mg/kg, intravenously, Q2W
  Interventions: Biological: HH-003 20mg/kg
- HH-003 3mg/kg (Experimental): HH-003 3mg/kg, intravenously, Q2W
  Interventions: Biological: HH-003 3mg/kg

INTERVENTIONS:
Biological: HH-003 20mg/kg — HH-003 20mg/kg Q2W intravenously for 24 weeks
  Arms: HH-003 20mg/kg
Biological: HH-003 3mg/kg — HH-003 3mg/kg Q2W intravenously for 24 weeks
  Arms: HH-003 3mg/kg

SUMMARY:
This is an open-label phase IIa study of HH-003 to evaluate its antiviral activity and safety in subjects with chronic hepatitis B and hepatitis D co-infection. HH-003 is a human monoclonal antibody targeting the pre-S1 domain of the HBV large envelope protein. It blocks engagement of preS1 with sodium taurocholate co-transporting polypeptide (NTCP), the cellular receptor for HBV/HDV.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form;
* Male or female subjects aged from 18 to 70 years inclusively;
* 18 kg/m2≤BMI≤32 kg/m2, body weight ≥45 kg for men and ≥40 kg for women;
* Positive HBsAg, anti-HDV IgG antibody and HDV RNA at screening;
* Women of childbearing potential or male subjects with female partners of childbearing potential should agree to use an adequate and highly effective contraceptions from screening to the end of study or until 12 weeks after last dose of the study drug (whichever is longer).

Exclusion Criteria:

* Be pregnant or lactating at screening;
* Subjects with decompensated liver cirrhosis;
* Subjects with liver dysfunction (including but not limited to ascites, hepatic encephalopathy and upper gastrointestinal bleeding) within 3 months prior to screening;
* Average daily alcohol consumption >40g for men and >20g for women or drug abuse within 6 months prior to screening;
* Subjects with other serious diseases that is inappropriate for study participation per the Investigator's or the Sponsor's discretion (including but not limited to serious cardiac or pulmonary disease, chronic or recurrent urinary disorders, uncontrolled diabetes and autoimmune diseases, epilepsy requiring treatment);
* History of hepatocellular carcinoma (HCC) or hepatocellular carcinoma suggested by liver histopathology or liver imaging;
* Interferon antiviral therapy within 1 year prior to screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with HBV DNA Negativation or Decrease by ≥1 log10 from Baseline at Week 24 | Week 24
Percentage of Participants with HDV RNA Negativation or Decrease by ≥1 log10 from Baseline at Week 24 | Week 24
Change from Baseline in Serum HBsAg Levels at Week 24 | from baseline to Week 24

SECONDARY OUTCOMES:
Percentage of participants with ALT normalization at week 24 | Week 24
Changes from Baseline in Serum HBsAg Levels during the Study Period | from baseline to Week 48
Changes from Baseline in Serum HBV RNA Levels during the Study Period | from baseline to Week 48
Changes from Baseline in Serum HBV DNA Levels during the Study Period | from baseline to Week 48
Changes from Baseline in Serum HDV RNA Levels during the Study Period | from baseline to Week 48
Changes from Baseline in Serum HBeAg Levels in HBeAg-positive Subjects at Screening | from baseline to Week 48

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China